CLINICAL TRIAL: NCT04863586
Title: Prevalence of Coronavirus Disease 2019 in People With Multiple Sclerosis Taking Disease Modifying Therapies in England
Brief Title: COVID-19 and Multiple Sclerosis Disease Modifying Therapies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20NS041
Record Dates: First submitted 2021-04-27; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Multiple Sclerosis
Keywords: Covid19; Multiple sclerosis; Disease modifying therapies
MeSH Terms: conditions — COVID-19; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tested positive for SARS-CoV-2: Eligible participants who have had a positive SARS-CoV-2 test will be included in the case group of the study.
- Not tested for SARS-CoV-2: A random sample of age, sex, and DMT matched people with MS who have not been tested for SARS-CoV-2 will be included in the control group of the study.

SUMMARY:
The COVID-19 pandemic is a major concern for people on long-term treatments that modify the immune system function. People with multiple sclerosis (pwMS) form a large group who receive such treatments called disease modifying therapies (DMTs). Several types of DMTs with different effects on the immune system are being used for multiple sclerosis (MS). In the absence of large-scale national studies, the risk of COVID-19 among pwMS on various DMTs has not been established.

A few physician-reported registry-based studies have suggested that anti-CD20 monoclonal antibodies, such as ocrelizumab and rituximab, used in the treatment of MS can increase the risk of COVID-19. However, in our community-based COVID-19 study of a large cohort of pwMS as part of the UK MS Register, we could not demonstrate an association between DMTs and susceptibility to COVID-19. Other studies have not found any relationship between DMTs and the outcome of COVID-19 among pwMS.

To our knowledge, UK is the only country in the world that collects national data on DMT use, providing us with the opportunity to investigate the impact of DMTs on COVID-19 susceptibility and severity in a large population of pwMS. In England, no DMT is being dispensed without prior approval and specialised commissioning by the national Health Services (NHS) England & NHS Improvement (NHSE/I). The scheme, currently implemented in over 100 NHS Trusts in England, ensures that treatment decisions are made in line with agreed commissioning policy and are evidence-based. NHSE/I also has access to Public Health England (PHE) held data on all people who have had a SARS-CoV-2 test. By identifying all pwMS on DMTs and all those who have had a test for coronavirus and collecting data on the clinical outcome of their COVID-19 from their local NHS hospitals, we would be able to establish the risk of COVID-19 and the risk of contracting the infection associated with different DMTs. The findings of the study will help MS clinical teams address the concerns of pwMS about taking DMTs during the COVID-19 pandemic and update their guidelines on the measures pwMS need to take during these unprecedented times.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Diagnosed with MS
* Received treatment with a DMT

Exclusion Criteria:

* Not fulfilling the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all people with MS taking DMTs in England.
Sampling Method: Probability Sample
Enrollment: 14240 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of testing positive for SARS-CoV-2 in people with MS taking DMTs | 6 months
  The number of people with MS taking DMTs who have tested positive for SARS-CoV-2 among all people with MS taking DMTs in England.

SECONDARY OUTCOMES:
Clinical outcomes of COVID-19 among people with MS taking DMTs | 6 months
  To determine the clinical outcomes of COVID-19 (e.g., severity of disease, death, and recovery) in people with MS taking DMTs in England
Risk of contracting COVID-19 associated with individual DMTs/other clinical and paraclinical factors | 6 months
  To assess the risk of contracting COVID-19 associated with individual DMTs and other clinical (e.g., physical disability and comorbidities) and paraclinical (e.g., white blood cell and lymphocyte counts, vitamin D levels) factors among people with MS taking DMTs in England
Association between clinical outcomes of COVID-19 and individual DMTs/other clinical and paraclinical factors | 6 months
  To assess the association between clinical outcomes of COVID-19 and individual DMTs or other clinical (e.g., physical disability and comorbidities) and paraclinical (e.g., white blood cell and lymphocyte counts, vitamin D levels) factors among people with MS taking DMTs in England

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, FRCP, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No